CLINICAL TRIAL: NCT05508867
Title: A Phase 2 Randomized Clinical Study of MK-4280A (Coformulated Favezelimab [MK-4280] Plus Pembrolizumab [MK-3475]) Versus Physician's Choice Chemotherapy in PD-(L)1-refractory, Relapsed or Refractory Classical Hodgkin Lymphoma (KEYFORM-008)
Brief Title: A Study of Coformulated Favezelimab/Pembrolizumab (MK-4280A) Versus Physician's Choice Chemotherapy in PD-(L)1-refractory, Relapsed or Refractory Classical Hodgkin Lymphoma (MK-4280A-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4280A-008; MK-4280A-008 (Other: MSD); 2023-503615-14-00 (Registry Identifier: EU CT); U1111-1287-5864 (Registry Identifier: UTN); 2022-000371-39 (EudraCT Number)
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hodgkin Lymphoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Hodgkin Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Bendamustine Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Favezelimab/Pembrolizumab (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) by intravenous (IV) infusion on Day 1, then every three weeks (Q3W), for up to 35 infusions.
  Interventions: Biological: favezelimab/pembrolizumab
- Chemotherapy (Bendamustine or Gemcitabine) (Active Comparator): Participants will receive physician's choice of EITHER bendamustine by IV infusion at a dose between 90 and 120 mg/m^2 on Day 1 and Day 2 of either a 3- or 4-week cycle for up to 6 cycles OR gemcitabine by IV infusion at a dose between 800 and 1200 mg/m^2 on Day 1 and Day 8 of a 3-week cycle for up to 6 cycles.
  Interventions: Drug: bendamustine; Drug: gemcitabine

INTERVENTIONS:
Biological: favezelimab/pembrolizumab — Coformulated favezelimab/pembrolizumab (800 mg/200 mg), IV infusion
  Other Names: MK-4820A
  Arms: Favezelimab/Pembrolizumab
Drug: bendamustine — IV infusion
  Other Names: BENDEKA®
  Arms: Chemotherapy (Bendamustine or Gemcitabine)
Drug: gemcitabine — IV infusion
  Other Names: GEMZAR®
  Arms: Chemotherapy (Bendamustine or Gemcitabine)

SUMMARY:
Researchers are looking for a way to treat classical Hodgkin lymphoma (cHL) that is relapsed (the cancer has come back after treatment) or refractory (current treatment has stopped working to slow or stop cancer growth). Researchers want to learn if people who receive coformulated favezelimab/pembrolizumab (MK-4280A) live longer without the cancer getting worse compared to those who receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of classical Hodgkin lymphoma (cHL) that is 2-fluorodeoxyglucose-avid (FDG-avid).
* Has relapsed (defined as disease progression after most recent therapy) or refractory (defined as failed to achieve CR or PR to most recent therapy) cHL and exhausted all available treatment options with known clinical benefit.
* Has progressed on treatment with an anti-PD-(L)1 monoclonal antibody (mAb) administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies.
* Submits an archival (≤5 years) or newly obtained tumor tissue sample which has not been previously irradiated.

Exclusion Criteria:

* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy.
* History of central nervous system (CNS) metastases or active CNS involvement.
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic treatment.
* History of hemophagocytic lymphohisticytosis.
* Has an active seizure disorder that is not well controlled.
* Has clinically significant (ie, active) cardiovascular disease.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received prior radiotherapy within 2 weeks of start of study intervention or radiation related toxicities requiring corticosteroids.
* Has not adequately recovered from major surgical procedure.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* History of human immunodeficiency virus (HIV).
* Has had an allogeneic hematopoietic stem cell or solid organ transplantation within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per Lugano Response Criteria as Assessed by investigator | Up to approximately 39 months
  PFS is defined as the time from randomization to the first documented disease progression per Lugano criteria 2014 as assessed by investigator or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 39 months
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) per Lugano Response Criteria as Assessed by investigator | Up to approximately 39 months
  ORR is defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) per Lugano criteria 2014 as assessed by investigator.
Duration of Response (DOR) per Lugano Response Criteria as Assessed by investigator | Up to approximately 39 months
  For participants who demonstrate CR or PR per Lugano criteria 2014 as assessed by investigator, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experienced At Least One Adverse Event (AE) | Up to approximately 25 months
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (105):
- United States (16):
  - The University of Arizona Cancer Center - North Campus ( Site 2216), Tucson, Arizona
  - UCLA Hematology/Oncology - Santa Monica ( Site 2208), Los Angeles, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA-Hematology and Medical Oncology ( Site, Torrance, California
  - Moffitt Cancer Center ( Site 2200), Tampa, Florida
  - University of Kentucky Chandler Medical Center ( Site 2201), Lexington, Kentucky
  - University of Maryland-Greenebaum Comprehensive Cancer Center ( Site 2210), Baltimore, Maryland
  - Johns Hopkins University-The Sidney Kimmel Comprehensive Cancer Center ( Site 2206), Baltimore, Maryland
  - University of Michigan ( Site 2215), Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 2222), Grand Rapids, Michigan
  - Rutgers Cancer Institute of New Jersey ( Site 2217), New Brunswick, New Jersey
  - Roswell Park Cancer Institute ( Site 2220), Buffalo, New York
  - University Hospitals Cleveland Medical Center ( Site 2214), Cleveland, Ohio
  - Cleveland Clinic-Taussig Cancer Center ( Site 2203), Cleveland, Ohio
  - AHN West Penn Hospital ( Site 2213), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center ( Site 2205), Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Center ( Site 2212), Seattle, Washington
- Argentina (2):
  - Hospital Aleman-oncohematologic diseases ( Site 2302), Buenos Aires
  - Fundacion Centro Oncologico de Integración Regional-Medical Oncology ( Site 2301), Mendoza
- Australia (4):
  - The Townsville Hospital ( Site 0006), Townsville, Queensland
  - Royal Adelaide Hospital ( Site 0005), Adelaide, South Australia
  - Western Health-Sunshine & Footscray Hospitals-Cancer Services-Cancer Research ( Site 0002), St Albans, Victoria
  - Royal Perth Hospital-Haematology ( Site 0004), Perth, Western Australia
- Belgium (2):
  - UZ Leuven-Hematology ( Site 0101), Leuven, Vlaams-Brabant
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi, Namur
- Brazil (2):
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 0202), Barretos, São Paulo
  - Hospital Paulistano-Americas Oncologia ( Site 0207), São Paulo
- Canada (4):
  - Cross Cancer Institute ( Site 0313), Edmonton, Alberta
  - Princess Margaret Cancer Centre ( Site 0310), Toronto, Ontario
  - Jewish General Hospital ( Site 0309), Montreal, Quebec
  - McGill University Health Centre ( Site 0314), Montreal, Quebec
- Chile (2):
  - FALP-UIDO ( Site 0400), Santiago, Region M. de Santiago
  - Clínica Inmunocel ( Site 0407), Santiago, Region M. de Santiago
- China (15):
  - Anhui Provincial Cancer Hospital ( Site 0501), Hefei, Anhui
  - Beijing Hospital ( Site 0514), Beijing, Beijing Municipality
  - Peking University Third Hospital-Hematology ( Site 0519), Beijing, Beijing Municipality
  - The First Affiliated hospital of Xiamen University ( Site 0512), Xiamen, Fujian
  - Sun Yat-sen University Cancer Center ( Site 0500), Guangzhou, Guangdong
  - Henan Cancer Hospital ( Site 0515), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0509), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 0513), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0503), Changsha, Hunan
  - The First Hospital of Jilin University-Hematology ( Site 0516), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 0520), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University-Head and Neck Oncology ( Site 0502), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital-lymphoma ( Site 0506), Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital ( Site 0510), Hangzhou, Zhejiang
  - Ningbo First Hospital ( Site 0518), Ningbo, Zhejiang
- Czechia (3):
  - Fakultní nemocnice Brno Bohunice-Interni hematologicka a onkologicka klinika ( Site 0901), Brno, Brno-mesto
  - Fakultni nemocnice Hradec Kralove-IV. interni hematologicka klinika ( Site 0902), Hradec Králové
  - Vseobecna fakultni nemocnice v Praze-I. Interní klinika - klinika hematologie ( Site 0903), Prague
- France (6):
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou-haematology ( Site 0707), Rennes, Brittany Region
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE ( Site 0706), Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren ( Site 0704), Limoges, Haute-Vienne
  - Institut Curie - site Saint-Cloud ( Site 0708), Saint-Cloud, Hauts-de-Seine
  - CENTRE LEON BERARD-Medical oncology ( Site 0703), Lyon, Rhone
  - HENRI MONDOR HOSPITAL ( Site 0702), Créteil, Seine-et-Marne
- Germany (7):
  - Klinikum Stuttgart - Katharinenhospital ( Site 0804), Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Ulm-Department of Internal Medicine III ( Site 0805), Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Koeln-Klinik I für Innere Medizin ( Site 0801), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 0807), Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus ( Site 0806), Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-University Cancer Center Early Clinical Trial Unit (, Dresden, Saxony
  - Universitätsklinikum Leipzig ( Site 0803), Leipzig, Saxony
- Israel (6):
  - Rambam Health Care Campus ( Site 1004), Haifa
  - Carmel Hospital ( Site 1007), Haifa
  - Hadassah Medical Center-Hemato-Oncology ( Site 1000), Jerusalem
  - Rabin Medical Center-Hemato-Oncology ( Site 1001), Petah Tikva
  - Sheba Medical Center-Hemato Oncology ( Site 1005), Ramat Gan
  - Sourasky Medical Center ( Site 1002), Tel Aviv
- Mexico (2):
  - Centro de Infusion Superare ( Site 2503), Mexico City, Mexico City
  - Unidad Médica Onco-hematológica ( Site 2507), Puebla City
- Poland (5):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie-Oncology Department ( Site 1406), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckieg-Klinika Hematologii, Nowotworów Krwi i, Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Kilinka Onkologii I Hematologii ( Site, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 1402), Gdansk, Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Hematologii i Transplantacji S, Kielce, Świętokrzyskie Voivodeship
- South Korea (5):
  - Pusan National University Hospital-Internal Medicine ( Site 1704), Busan, Pusan-Kwangyokshi
  - Seoul National University Hospital ( Site 1701), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 1702), Seoul
  - Asan Medical Center-Department of Oncology ( Site 1703), Seoul
  - Samsung Medical Center ( Site 1700), Seoul
- Spain (8):
  - Hospital Universitario Marqués de Valdecilla ( Site 1805), Santander, Cantabria
  - Hospital Universitari Vall d'Hebron ( Site 1803), Barcelona, Catalonia
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 1812), A Coruña, La Coruna
  - Hospital Insular de Gran Canaria-Oncology ( Site 1807), Las Palmas de Gran Canaria, Las Palmas
  - Hospital General Universitario de Alicante ( Site 1806), Alicante
  - Hospital Universitario 12 de Octubre-Hemathology and hemotherapy ( Site 1810), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 1808), Málaga
  - Hospital Universitario de Salamanca - Complejo Asistencial U-Servicio de Hematologia ( Site 1801), Salamanca
- Sweden (2):
  - Skånes Universitetssjukhus Lund ( Site 1901), Lund, Skåne County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 1900), Uppsala, Uppsala County
- Ospedale Regionale Bellinzona e Valli-IOSI ( Site 1600), Bellinzona, Canton Ticino, Switzerland
- Turkey (Türkiye) (6):
  - Mega Medipol-Hematology ( Site 2005), Stanbul, Istanbul
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 2000), Ankara
  - Hacettepe Universite Hastaneleri-Department of Hematology ( Site 2006), Ankara
  - Antalya Egitim ve Arastırma Hastanesi ( Site 2011), Antalya
  - Ege Universitesi Hastanesi ( Site 2001), Izmir
  - Kocaeli Üniversitesi-Hematology ( Site 2009), Kocaeli
- United Kingdom (7):
  - Derriford Hospital ( Site 2107), Plymouth, Devon
  - The Beatson West of Scotland Cancer Centre ( Site 2110), Glasgow, Glasgow City
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 2105), London, London, City of
  - GenesisCare - Oxford ( Site 2104), Oxford, Oxfordshire
  - St James's University Hospital ( Site 2109), Leeds
  - Leicester Royal Infirmary ( Site 2100), Leicester
  - Clatterbridge Cancer Centre - Liverpool-Heamatology ( Site 2108), Liverpool

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26284&tenant=MT_MSD_9011